CLINICAL TRIAL: NCT05183373
Title: Inflammation and Clotting Abnormalities in Aneurysmal Coronary Artery Disease
Acronym: CARE-ANUERYSM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: John Paul II Hospital, Krakow (Other)
Collaborators: Jagiellonian University (Other); National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/39/NZ5/02863
Record Dates: First submitted 2022-01-05; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Aneurysm; Abdominal Aortic Aneurysm; Coronary Disease
Keywords: Coronary Artery Aneurysm; Inflammation; Fibrin Clot Lysis Time; Coronary Disease; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Coronary Aneurysm; Aortic Aneurysm, Abdominal; Coronary Disease; Inflammation | interventions — Bleeding Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aneurysmal coronary artery disease: Patients with coronary artery ectasia or/and aneurysm diagnosed during coronary angiography
  Interventions: Other: Evaluation of inflammation and clotting
- Abdominal aortic aneurysm: Patients with diagnosed with abdominal aortic aneurysm
  Interventions: Other: Evaluation of inflammation and clotting
- Coronary artery disease: Patients with diagnosed with coronary artery disease
  Interventions: Other: Evaluation of inflammation and clotting

INTERVENTIONS:
Other: Evaluation of inflammation and clotting — Evaluation of inflammation biomarkers (such as 8-isoprostane, Il-6) and fibrin clot properties (such as clot lysis time, clot permeability)

SUMMARY:
The main objective of the CARE-ANEURYSM project is to evaluate inflammation and clotting abnormalities in patients with aneurysmal coronary artery disease in relation to patients with abdominal aortic aneurysm or coronary artery disease (acting as controls).

DETAILED DESCRIPTION:
The trial will enrol 180 patients, 60 in each of three groups: 1) aneurysmal coronary artery disease; 2) abdominal aortic aneurysm; 3) coronary artery disease. In addition, up to 250 patients with aneurysmal coronary disease will be follow for clinical outcomes in relation to controls (prognosis group).

The primary research question of this project is to evaluate wheter the inflammation and clotting abnormalities in patients with aneurysmal coronary artery disease differ from ones in abdominal aortic aneurysm or coronary artery diseases. Study endpoints include the level of inflammation biomarkers and fibrin clot properties in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years old
* Angiographically confirmed coronary artery ectasia or aneurysm (Arm I)
* Abdominal aortic aneurysm (Arm II)
* Angiographically confirmed coronary artery disease (Arm III)

Exclusion Criteria:

* Less than 12 months from ACS
* Actual oral anticoagulant therapy
* Actual antiplatelet therapy other than aspirin
* Heart failure NYHA IV
* Untreated hyperthyroidism or hypothyroidism
* Severe comorbidities
* Lack of consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comer, consecutive patients with the contiontds under the evaluation in this study will be screen for enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Inflammation | Baseline (at enrolment)
  Level of inflammation biomarkers (such as 8-isoprostane, Il-6) in each group
Clotting | Baseline (at enrolment)
  Fibrin clot properties (such as clot lysis time, clot permeability) in each group
Composite Clinical outcome after 1 year | 1 year after the enrolment
  Death, stroke, myocardial infarction
Composite Clinical outcome after 5 years | 5 years after the enrolment
  Death, stroke, myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musiałek, MD, DPhil, Principal Investigator — John Paul II Hospital, Krakow
Locations (1):
- Department of Cardiac and Vascular Diseases, John Paul II Hospital, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doi T, Kataoka Y, Noguchi T, Shibata T, Nakashima T, Kawakami S, Nakao K, Fujino M, Nagai T, Kanaya T, Tahara Y, Asaumi Y, Tsuda E, Nakai M, Nishimura K, Anzai T, Kusano K, Shimokawa H, Goto Y, Yasuda S. Coronary Artery Ectasia Predicts Future Cardiac Events in Patients With Acute Myocardial Infarction. Arterioscler Thromb Vasc Biol. 2017 Dec;37(12):2350-2355. doi: 10.1161/ATVBAHA.117.309683. Epub 2017 Oct 19. PMID 29051141
- [Background] Kawsara A, Nunez Gil IJ, Alqahtani F, Moreland J, Rihal CS, Alkhouli M. Management of Coronary Artery Aneurysms. JACC Cardiovasc Interv. 2018 Jul 9;11(13):1211-1223. doi: 10.1016/j.jcin.2018.02.041. PMID 29976357
- [Background] Gunasekaran P, Stanojevic D, Drees T, Fritzlen J, Haghnegahdar M, McCullough M, Barua R, Mehta A, Hockstad E, Wiley M, Earnest M, Tadros P, Genton R, Gupta K. Prognostic significance, angiographic characteristics and impact of antithrombotic and anticoagulant therapy on outcomes in high versus low grade coronary artery ectasia: A long-term follow-up study. Catheter Cardiovasc Interv. 2019 Jun 1;93(7):1219-1227. doi: 10.1002/ccd.27929. Epub 2018 Nov 4. PMID 30393992
- [Background] Boles U, Johansson A, Wiklund U, Sharif Z, David S, McGrory S, Henein MY. Cytokine Disturbances in Coronary Artery Ectasia Do Not Support Atherosclerosis Pathogenesis. Int J Mol Sci. 2018 Jan 16;19(1):260. doi: 10.3390/ijms19010260. PMID 29337902
- [Background] Brunetti ND, Salvemini G, Cuculo A, Ruggiero A, De Gennaro L, Gaglione A, Di Biase M. Coronary artery ectasia is related to coronary slow flow and inflammatory activation. Atherosclerosis. 2014 Apr;233(2):636-640. doi: 10.1016/j.atherosclerosis.2014.01.018. Epub 2014 Jan 28. PMID 24553454
- [Derived] Chmiel J, Natorska J, Zabczyk M, Musialek P. Fibrin clot properties in coronary artery ectatic disease: Pilot data from the CARE-ANEURYSM Study. Kardiol Pol. 2023;81(11):1145-1148. doi: 10.33963/v.kp.96983. Epub 2023 Sep 3. No abstract available. PMID 37660376